CLINICAL TRIAL: NCT01451372
Title: Routine Use of Sensor-Augmented Pump Therapy - a Follow up Study
Status: Completed | Type: Observational
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Other Study IDs: SW01
Record Dates: First submitted 2011-09-29; First posted 2011-10-13 (Estimated); Results first posted 2019-02-27 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2018-10

CONDITIONS: Diabetes
Keywords: Diabetes; CGM; CSII
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of this study is to document the routine practice in continuous glucose monitoring (CGM) in patients treated with sensor-augmented pump therapy and to assess clinical outcome (HbA1c) before the start of the sensor use to the end of the follow-up period. Moreover, data on treatment satisfaction, and fear of hypoglycemia, cost of the therapy, side effects and treatment interruption will be collected.

DETAILED DESCRIPTION:
The most advanced technologies for the treatment of type 1 diabetes mellitus (T1DM) include insulin pumps for continuous subcutaneous insulin infusion (CSII) and glucose sensors allowing continuous glucose monitoring(CGM). Randomized controlled trials have shown that access to CGM can improve control in poorly-controlled patients regardless of insulin treatment therapy via reduced hyper- and hypoglycaemic excursions and improved mean HbA1c value.

The Medtronic personal CGM device is composed of a glucose sensor linked to a MiniLink REAL-Time Transmitter, which transmits data from the glucose sensor to the insulin pump. The integration of these two technologies (CSII and personal CGM) into one system is called sensor-augmented pump therapy (SAP).The devices are CE-marked and routinely used in clinical practice in the Swedish market.

Based on the clinical evidences provided, the Swedish Dental and Pharmaceutical Benefits Agency (TLV) concluded that the personal CGM when used in combination to a Medtronic insulin pump as SAP should be included in the Swedish reimbursement system. However the decision was upon specific patient indications:

Patients with two or more severe hypoglycemias/year that require help from another person or Patients with HbA1c of at least 9%, in cases where optimized insulin therapy has not been effective or Children taking at least 10 medically required plasma glucose tests (fingersticks) per 24 hours and that certain follow-up information has to be complemented and submitted to TLV before March 1st, 2012.

TLV requires follow-up information on T1 diabetes patients using SAP in Swedish clinical practice and based on the following outcome parameters:

HbA1c-level of the patients Quality of life with use of CGM Side effects and therapy interruptions. Use and costs of the therapy Frequency of hypoglycemia Therefore, this project will observe the routine practice of personal CGM utilization in combination to Medtronic insulin pumps in T1DM patients in Sweden in approximately 15 investigational centers.

The aim of this project is to reflect the daily practice in personal CGM therapy (sensor and MiniLink REAL-Time Transmitter) usage in diabetes patients treated with Medtronic insulin pumps in Sweden. Data on the HbA1c value before and up to six months use of personal CGM will be collected and information on the outcomes requested by TLV will be included in the study. The patient reported outcomes will be supplemented with patient preference data and will be estimated with a willingness-to-pay (WTP) approach.

ELIGIBILITY:
Inclusion Criteria:

* Patient (and/or legal representative) has signed Patient Informed Consent(PIC) AND
* Patient (0-69 years) was diagnosed with Type 1 DM and has been on insulin pump therapy (without any additional insulin injection) for at least 3 months prior to signature of the PIC AND
* HbA1c ≥ 7 %) or
* has experienced at least 2 severe hypoglycemic events in the last 12 months or
* is performing on average more than 10 SMBG per day AND The patient has used, or is using or will start using continuous glucose monitoring as part of the CSII therapy for at least 70% of the time for a minimum of 3 months.

Exclusion Criteria:

* Participation in any other clinical trial - currently and/or in the last 3 months prior signature of informed consent and/or during the retrospective period of data collection.
* Unwillingness to perform at least 4 BG tests per day
* Unwillingness to maintain contact with HCP
* For children: no reliable contact person
* PREGNANT woman and wish of pregnancy
* Vision and hearing impairment not allowing pump use
* Any disease or drug treatment that can interfere with the outcome of sensor usage.

Max Age: 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Population will be selected from Primary Care Clinics.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2011-06; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Örtqvist, MD, Principal Investigator — ALB, Karolinska Universitetssjukhuset Solna
Locations (1):
- Medtronic AB, Stockholm, Kista, Sweden

RESULTS

PARTICIPANT FLOW:
Groups:
- Type 1 Diabetes Subjects Using CGM: Type 1 Diabetes Subjects using CGM in Sweden
Period: Overall Study
Arm/Group | Type 1 Diabetes Subjects Using CGM
Started | 69
Completed | 69
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Type 1 Diabetes Subjects Using CGM
Number analyzed (Participants) | 69
Age, Customized [Mean (Full Range); unit: years]
  Age, Continuous | 33 [3 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 22
Region of Enrollment [Number; unit: participants]
  Sweden | 69

OUTCOME MEASURES:

1. Primary Outcome: Daily Usage of Blood Glucose Test (BG Testing)
Description: Daily usage of blood glucose test 0-24 months after CGM usage. This information is collected in a journal questionnaire
Time Frame: 24 months
Population: journal questionnaires about blood glucose testing were collected from 65 out of 69 subjects
Measure: Mean (Standard Deviation); unit: number of blood glucose test per day
Arm/Group | Type 1 Diabetes Subjects Using CGM
Number analyzed (Participants) | 65
number of blood glucose test per day | 4.35 (2.4)

2. Secondary Outcome: Frequency of Sensor Usage Per Month
Description: Frequency of sensor usage per month during the study. This information is collected in a journal questionnaire
Time Frame: 24 months
Population: Journal questionnaires about sensor usage were collected from 61 out of 69 subjects
Measure: Mean (Standard Deviation); unit: number of sensor used per month
Arm/Group | Type 1 Diabetes Subjects Using CGM
Number analyzed (Participants) | 61
number of sensor used per month | 4 (1.5)

ADVERSE EVENTS:
Time Frame: 24 month
Arm/Group | Type 1 Diabetes Subjects Using CGM
All-Cause Mortality (participants affected / at risk) | 18/69
Serious Adverse Events (participants affected / at risk) | 0/69
Other Adverse Events (participants affected / at risk) | 18/69
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Type 1 Diabetes Subjects Using CGM (N=69)
Infection (Infections and infestations) | 5 (5)
Skin Irritation (Skin and subcutaneous tissue disorders) | 15 (15)
Inflammation (Immune system disorders) | 3 (3)
Bleeding (Injury, poisoning and procedural complications) | 1 (1)
Other (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days